CLINICAL TRIAL: NCT04639115
Title: A Phase 1, Multicenter, Open-Label Study to Evaluate the Effect of Mild or Moderate Hepatic Impairment on the Multiple-Dose Pharmacokinetics of Ozanimod
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RPC-1063-CP-004; U1111-1257-6851 (Registry Identifier: WHO)
Record Dates: First submitted 2020-11-17; First posted 2020-11-20 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Liver Diseases; Digestive System Diseases
Keywords: Mild and moderate Hepatic impairment; Healthy volunteer; Ozanimod
MeSH Terms: conditions — Liver Diseases; Digestive System Diseases; Lymphoma, Follicular | interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ozanimod in subjects with mild hepatic impairment (Experimental): Participants will receive ozanimod 0.23 mg once daily (QD) on Days 1 to 4, 0.46 mg QD on Days 5 to 7, and 0.92 mg QD on Day 8 in subjects with mild hepatic impairment
  Interventions: Drug: Ozanimod
- Ozanimod in subjects with moderate hepatic impairment (Experimental): Participants will receive ozanimod 0.23 mg once daily (QD) on Days 1 to 4, 0.46 mg QD on Days 5 to 7, and 0.92 mg QD on Day 8 in subjects with moderate hepatic impairment
  Interventions: Drug: Ozanimod
- Ozanimod in healthy subjects (Experimental): Participants will receive ozanimod 0.23 mg once daily (QD) on Days 1 to 4, 0.46 mg QD on Days 5 to 7, and 0.92 mg QD on Day 8 in healthy subjects
  Interventions: Drug: Ozanimod

INTERVENTIONS:
Drug: Ozanimod — Ozanimod
  Other Names: RPC-1063, Zeposia

SUMMARY:
This is a Phase 1, multicenter, nonrandomized, open-label, parallel-group study in participants with mild or moderate hepatic impairment, and in participants with normal hepatic function.

Degrees of hepatic impairment will be determined during screening by the participant's score according to Pugh's Modification of Child's Classification of Severity of Liver Disease.

Participants will be enrolled in Groups 1 through 3 as follows:

* Group 1 (mild hepatic impairment): A total of approximately 8 participants with a Child-Pugh score of 5 to 6.
* Group 2 (moderate hepatic impairment): A total of approximately 8 participants with a Child-Pugh score of 7 to 9.
* Group 3 (normal hepatic function): Approximately 8 to 16 participants will be matched to Participants in Groups 1 and 2. Normal hepatic function participants are allowed to match multiple hepatic impairment participants. Participants will be matched by sex, age (± 10 years), weight (± 20%), and smoking status.

ELIGIBILITY:
Inclusion Criteria:

Acceptable methods of birth control in this study are the following:

* Combined hormonal (oestrogen and progestogen containing) contraception, which may be oral, intravaginal, or transdermal
* Progestogen-only hormonal contraception associated with inhibition of ovulation, which may be oral, injectable, or implantable
* Placement of an intrauterine device or intrauterine hormone-releasing system
* Bilateral tubal occlusion
* Vasectomized partner
* Complete sexual abstinence

All participants:

Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not acceptable methods of contraception.

Inclusion Criteria for Participants with Mild or Moderate Hepatic Impairment (Groups 1 and 2)

Each participant with mild or moderate hepatic impairment must satisfy the following criteria to be enrolled in the study:

* Participant has mild (5 to 6 points) or moderate (7 to 9 points) hepatic impairment per the Child-Pugh system (Appendix B).
* Participant should be enrolled into the group corresponding to the Child-Pugh classification score that most accurately reflects the most severe hepatic disease classification within the past 6 months of signing the ICF (based on past medical history or PE observation).
* If a Child-Pugh score was previously calculated and documented in the last 6 months, and it is more severe than the one calculated at Screening, then that previous value will be used for study entry purposes. If the Screening Child-Pugh score is more severe, then it will be used. If no score was calculated in the 6 months prior to Screening, then the score obtained at Screening will be used. Adequate documentation should be provided to substantiate the Child-Pugh score assigned to each participant.
* Participant must be medically stable for at least 4 weeks before Screening with clinically acceptable medical history (eg, no worsening of clinical signs of hepatic impairment, or no worsening of total bilirubin or prothrombin time by more than 50%), PE, clinical laboratory tests, vital signs, and 12-lead ECGs consistent with the underlying stable hepatic impairment condition, as judged by the Investigator.
* Participant with laboratory parameters that are considered clinically significant beyond those consistent with their degree of hepatic impairment may be included if, in the opinion of the Investigator and Medical Monitor, these findings will not interfere with the study or introduce additional safety risk to the participant.
* Participant must be stable on a concomitant medication and/or treatment regimen (defined as not starting a new treatment/medication[s] or a change in the dosage or frequency of the concomitant medication[s] within 2 weeks before dosing with ozanimod).
* Participant must have estimated creatinine clearance ≥ 50 mL/min at Screening as calculated by the Cockcroft-Gault formula.

Inclusion Criteria for Matched Normal Hepatic Function Participants (Group 3)

Each matched participant must satisfy the following criteria to be enrolled in the study:

* Participant is in good health as determined by past medical history, PE, vital signs, ECG, and clinical laboratory safety tests. Clinical laboratory safety tests (ie, hematology, coagulation, chemistry, and urinalysis) must be within normal limits or clinically acceptable as judged by the Investigator.
* Participant must match a participant in Groups 1 and/or 2, with respect to sex, age (± 10 years), weight (± 20%) and smoking status. One normal hepatic function participant can be matched to 2 hepatic impairment participants (one in Group 1 and one in Group 2), but no more than one hepatic impairment participant in the same group.

Exclusion Criteria:

Exclusion Criteria for All Participants

The presence of any of the following will exclude a participant from enrollment:

* Participant has any condition including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study.
* Participant has any condition that confounds the ability to interpret data from the study.
* Participant has a seated blood pressure outside 90 to 155 mmHg systolic or 50 to 95 mmHg diastolic at Screening or Day -1.
* Participant has a seated pulse rate outside 55 to 90 beats per minute (bpm) at Screening or Day -1.
* Participant has a positive serum test for human immunodeficiency virus (HIV) at Screening or Day -1.
* Participant with any active infection including hepatitis.
* Participant has a positive alcohol urine or breath test at Screening or Day -1.
* Participant has received any investigational drug within 30 days or 5 times the elimination half-life (if known), whichever is longer, prior to the first dose of IP.
* Participant has consumed pomelo-variety citrus fruits or juice (including pomelo, grapefruit, Seville oranges) within 7 days prior to the first dose of IP or herbal supplements including St. John's wort within 28 days prior to the first dose of IP.
* Participant fails or is unwilling to abstain from strenuous physical activities for at least 24 hours prior to the first dose of IP.
* Participant has poor peripheral venous access.
* Participant has donated greater than 400 mL of blood within 60 days prior to Day 1.
* Participant has history of hypersensitivity or allergic reaction to S1P receptor modulators.
* Participant has used any of the following systemic medications:

  1. Strong inhibitors of CYP3A, and all inhibitors of CYP2C8 or BCRP, (ie, cyclosporine, eltrombopag, gefitinib) within 7 days or 5 half-lives, whichever is longer, prior to Day 1, or
  2. Strong inducers of CYP3A, and all inducers of CYP2C8 within 14 days or 5 halflives, whichever is longer, prior to Day 1, or
  3. Any known MAO inhibitors within 30 days or 5 half-lives, whichever is longer, prior to Day 1. Examples of MAO inhibitors include but are not limited to phenelzine, selegiline, isocarboxazid, rasagiline, tranylcypromine, pargyline, procarbazine, and furazolidone.
* Participant who in the last 6 months of signing the ICF experienced myocardial infarction, unstable angina, stroke, transient ischaemic attack, decompensated heart failure requiringmhospitalization or New York Heart Association (NYHA) Class III/IV heart failure.
* Participant with history or presence of second-degree atrioventricular (AV) block Type II or third-degree AV block or sick sinus syndrome unless the patient has a functioning pacemaker.
* Participant with history of cardiac arrest, cerebrovascular disease, uncontrolled hypertension, or severe untreated sleep apnoea, history of recurrent syncope or symptomatic bradycardia
* Participant with pre-existing significant QT interval prolongation (QTc greater than 500 msec) or other risks for QT prolongation, and patients on medicinal products other than beta-blockers and calcium-channel blockers that may potentiate bradycardia.
* Participant on class Ia (eg, quinidine, disopyramide) or class III (eg, amiodarone, sotalol) antiarrhythmic medicinal products, which have been associated with cases of torsades de pointes in patients with bradycardia have not been studied with ozanimod.

Exclusion Criteria for Participants with Hepatic Impairment (Groups 1 and 2)

The presence of any of the following will exclude a hepatically-impaired participant from enrollment:

* Participant has any serious medical condition (excluding hepatic impairment and related complications), clinically significant laboratory abnormality not related to hepatic impairment and related complications, or psychiatric illness that would prevent the participant from participating in the study per Investigator discretion.
* Participant has current hepatic encephalopathy with time-or place-disorientation, somnolence, stupor, coma, no personality/behavior, rigidity, or hyperactive reflexes - or has had such within 1 month of Screening.
* Participant has planned liver transplantation within 6 months of Screening or has received a liver transplant, transjugular intrahepatic portosystemic shunt, or transjugular intrahepatic portosystemic stent shunting procedure.
* Participant has a history of alcoholism, drug abuse, or addiction within 6 months prior to Screening.
* Participant has a positive urine drug screen including cotinine (non-smokers and former smokers only) (except for prescribed medications such as benzodiazepines) at Screening or Day -1. Tetrahydrocannabinol use (as permitted by local law) is not allowed within 14 days prior to Day 1 and during the study.
* Participant has any history of cholecystectomy, clinically significant cardiovascular or cerebrovascular disease.
* Participant has severe ascites at Screening or Day -1.
* Participant has hepatocellular carcinoma or acute liver disease (eg, caused by an infection or drug toxicity).
* Participant chronically or routinely uses more than 2 g of acetaminophen daily.

Exclusion Criteria for Matched Normal Hepatic Function Participants (Group 3)

The presence of any of the following will exclude a matched normal hepatic function participant from enrollment:

* Participant has any significant medical condition or psychiatric illness that would prevent the participant from participating in the study (as determined by the Investigator).
* Participant has a history of alcoholism, drug abuse, or addition within 24 months prior to Screening.
* Participant has a positive test result for hepatitis B surface antigen and/or hepatitis C antibody.
* Participant has a positive urine drug test (except for cotinine in smokers) at Screening or Day -1.
* Participant has used any systemic over-the-counter medication (excluding acetaminophen up to 2 g/day and low dose aspirin) within 7 days prior to Day 1, or any systemic prescription medication (except for contraceptives) within 28 days or 5-half-lives, whichever is longer, prior to Day 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - AUClast on Day 8 (Ozanimod, CC112273 and CC1084037) | Up to day 8
  AUC from time zero to the last measured time point
Pharmacokinetics - AUC∞ on Day 8 (Ozanimod, CC112273 and CC1084037) | Up to day 8
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacokinetics - Cmax on Day 8 (Ozanimod, CC112273 and CC1084037) | Up to day 8
  Maximum observed plasma concentration
Pharmacokinetics - Cmin on Day 8 (Ozanimod, CC112273 and CC1084037) | Up to day 8
  Minimum observed plasma concentration
Pharmacokinetics - AUCtau on Day 8 (Ozanimod, CC112273 and CC1084037) | Up to day 8
  Area under the plasma concentration-time curve from time zero to dosing interval

SECONDARY OUTCOMES:
Adverse Events (AEs) | From the time the ICF is signed until 64 ± 3 days after the last dose of ozanimod treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a Participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the Participant's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE
Pharmacokinetics -Cmax on Days 1 and 5 (Ozanimod, CC112273 and CC1084037) | Days 1 and 5
  Maximum observed plasma concentration
Pharmacokinetics -Cmin on Days 1 and 5 (Ozanimod, CC112273 and CC1084037) | Days 1, and 5
  Minimum observed plasma concentration
Pharmacokinetics - AUCtau on Days 1 and 5 (Ozanimod, CC112273 and CC1084037) | Days 1 and 5
  Area under the plasma concentration-time curve from time zero to dosing interval
Pharmacokinetics - Tmax (Ozanimod, CC112273 and CC1084037) | Days 1, 5, and 8
  Time to reach maximum observed plasma concentration
Pharmacokinetics - AUClast (Ozanimod, CC112273 and CC1084037) | From Day 8 till Day 72
  AUC from time zero to the last measured time point
Pharmacokinetics - t1/2 (Ozanimod, CC112273 and CC1084037) | From Day 8 till Day 72
  Terminal elimination half-life
Pharmacokinetics - Vz/F (Ozanimod) | From Day 8 till Day 72
  Apparent volume of distribution when dosed orally
Pharmacokinetics - CL/F (Ozanimod) | From Day 8 till Day 72
  Apparent total plasma clearance when dosed orally
Pharmacokinetics - fu (Ozanimod, CC112273 and CC1084037) | Day 1 and Day 8
  Unbound fraction
Pharmacokinetics - Cmax,u (Ozanimod, CC112273 and CC1084037) | Days 1, 5, and 8
  Maximum observed plasma concentration
Pharmacokinetics - AUC∞,u (Ozanimod, CC112273 and CC1084037) | From Day 8 till Day 72
  Unbound AUC∞
Pharmacokinetics - AUClast,u (Ozanimod, CC112273 and CC1084037) | From Day 8 till Day 72
  Unbound AUClast
Pharmacokinetics - AUCtau,u (Ozanimod, CC112273 and CC1084037) | Days 1, 5, and 8
  Unbound AUCtau
Pharmacokinetics - M/P AUCtau ratio (CC112273 and CC1084037) | Days 1, 5, and 8
  Molecular weight corrected metabolite-to-parent AUC from time zero to dosing interval ratio

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - University of Miami Miller School of Medicine, Miami, Florida
  - Orlando Clinical Research Center OCRC, Orlando, Florida
  - The Texas Liver Institute, San Antonio, Texas

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com